CLINICAL TRIAL: NCT06974227
Title: Validation Study of an Assistive Pulse Data Collection Device
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Logistics and Supply Chain MultiTech R&D Centre, Hong Kong (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PRM
Record Dates: First submitted 2025-03-09; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-03

CONDITIONS: Healthy Male and Female Subjects
Keywords: machine; pulse; wave form; TCM

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Assistive Pulse Data Collection (APDC) Device (Experimental): An Assistive Pulse Data Collection Device prototype has been designed and manufactured by the Logistics and Supply Chain MultiTech R&D Centre, Hong Kong. The device comprises a pulse sensor to record the patient's pulse and digitalize the pulse feature into waveform data. The digitalized waveform data is then converted the electronic signal into mechanical vibration that responds to the patient's pulse.
  Interventions: Device: Assistive Pulse Data Collection (APDC) Device

INTERVENTIONS:
Device: Assistive Pulse Data Collection (APDC) Device — An Assistive Pulse Data Collection Device prototype has been designed and manufactured by the Logistics and Supply Chain MultiTech R&D Centre, Hong Kong. The device comprises a pulse sensor to record the patient's pulse and digitalize the pulse feature into waveform data. The digitalized waveform data is then converted the electronic signal into mechanical vibration that responds to the patient's pulse.

SUMMARY:
Background: Traditional Chinese Medicine (TCM) relies on pulse diagnosis, a subjective and complex method that is crucial for assessing patients' health status. The COVID-19 pandemic has disrupted healthcare delivery, highlighting the need for remote diagnostic tools. To address this, an Assistive Pulse Data Collection Device (APDC) has been developed to capture and regenerate pulse features for remote pulse assessment in TCM.

Objective: This study aims to validate the accuracy and reliability of the APDC by assessing its agreement with Chinese Medicine Practitioners (CMPs) and collecting users' feedback.

Intervention: The APDC consists of a radial artery viewing device, pulse collection device, and pulse regeneration device.

Methods: Subjects will be recruited via social media and posters at the University. Inclusion criteria include age 18-65 years and BMI 18.5-22.5 kg/m2, while exclusion criteria include a dorsally located radial artery. Registered CMPs with at least 5 years of clinical experience will assess the pulse from both participants and the regenerated pulse by the device.

Outcome Assessment: Agreement in pulse features between the subjects' real pulse and the pulse regeneration device will be assessed using a self-developed questionnaire, covering frequency, rhythm, wideness, and force. Quantitative and qualitative feedback from subjects and CMPs will be collected to assess their views on the APDC Device in terms of satisfaction, ease of use, and comfortability.

DETAILED DESCRIPTION:
This study aims to assess whether the CMP can correctly recognize the pulse feature generated from the APDC Device and match it with the subjects. Its purpose is to ensure that the device-regenerated pulse resembles the subjects' pulse.

Feasibility Phase During the Feasibility Phase, users' experience from both CMPs and subjects will be collected for the team to refine the setting of the APDC Device.

Procedure

1. A subject's pulse features will be recorded by the APDC Device;
2. Three CMPs will assess the subject's pulse of both hands and then the regeneration pulse from the APDC Device;
3. The CMPs will rate the agreement, using a predefined record form (appendix 1), on the likeliness between the subjects' pulse and PTSE-regenerated pulse, in the respects of frequency, rhythm, wideness, and force (5-point Likert for each domain, from "Strongly disagree" to "strongly agree")
4. Subjects' user experience will be assessed by a questionnaire (appendix 2);
5. The above steps repeat until 10 subjects' pulses have been assessed.

The engineer team will then adjust and improve the machine based on the user feedback.

Pilot Phase In the Pilot Phase, the above procedure will be repeated until 12 CMPs' and 35 subjects' feedback have been collected.

Blinding the practitioners is not feasible due to the inherent differences between the simulator and a real subject. In this case, the study design focuses on the practitioners' ability to match the pulse features from the simulator to those of the patients using categorical responses.

Procedure

1. Three CMPs will take turns to assess five subjects' pulses;
2. The CMPs will categorize each subject's pulse, in the respects of frequency, rhythm, wideness, and force at three places of the wrist, which are known as cun, guan, and chi;
3. The CMPs will then assess the five regenerated pulses from the APDC Device in random order. They will be informed that the pulses are generated from the five subjects they have just assessed in random order;
4. The CMPs will categorize and the APDC-regenerated pulse, using the same approach; they will be asked to match the PTSE-regenerated pulse with the subjects.
5. The above procedure will repeat until thirty subjects are assessed.

Subject recruitment Subjects will be recruited via social media and posters at the University. All subjects will be required to sign a consent form indicating their voluntary participation. Their socio-demographic characteristics will be recruited. The Pulse Taking System Device will digitalize the pulse feature in waveform data. Registered CMPs with at least 5 years of clinical experience will be recruited to assess the pulse from both participants and the device; afterward, they will fill out a predefined record form to rate the pulse characteristics. A HK$100 supermarket coupon will be given to the subject as an incentive upon completion of either phase 1 or 2.

Subjects

* Inclusion criteria

  1. Age 18-65 years
  2. BMI 18.5-22.5 kg/m2
  3. Willing to give informed consent
* Exclusion criteria 1. dorsally located radial artery

Pulse taking setting The CMPs will assess the subjects' pulse as if they were in clinical practice. Subjects will sit on a chair, put their arm on a table, and position their wrist on a pulse pillow. The CMP will assess the subjects' pulse for up to one minute each.

Outcome assessment Agreement in pulse feature between the CMPs and the pulse regeneration device will be assessed using a self-developed questionnaire. The questionnaire will cover the pulse features including frequency, rhythm, wideness, and force.

Users' experience As the APDC Device consists of three parts, namely artery viewing device, pulse collection device, and pulse re-generation device. Device will be assessed separately.

Quantitative feedback from the subjects and CMPs will be collected via a self-developed questionnaire using 5-point Likert items to assess their view on the Pulse Taking System Device, in terms of the satisfaction, ease to use, and comfortability etc.

Qualitative feedback from the subjects and CMPs will be collected using open end questions by a self-completed questionnaire. The ease of use and further suggestions for the pulse taking system device will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years
2. BMI 18.5-22.5 kg/m2
3. Willing to give informed consent

Exclusion Criteria:

1. dorsally located radial artery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Rating on the Agreement in pulse feature | Baseline
  CMPs will rate their level of agreement with statements regarding the similarity between the machine-generated pulse and the actual pulse of subjects. Responses will be recorded using a 5-point Likert scale, ranging from 1 (Strongly Disagree) to 5 (Strongly Agree). The questionnaire (4-item) evaluated four key pulse attributes: frequency, rhythm, wideness, and force.
  CMPs will assess the extent to which they agreed that the frequency of the machine-regenerated pulse accurately resembled that of a real person's pulse. Similarly, they evaluated the rhythm, wideness, and force of the machine-generated pulse in comparison to the actual pulse.

SECONDARY OUTCOMES:
Subjects feedback on the device | Baseline
  Subjects' feedback on their experience with the pulse measurement process was collected. Subjects will indicate their level of agreement with various statements using a 5-point scale (1 "Not at all" to 5 "Very Much"). The questionnaire is 4-item, each focused on four key areas: comfort during the measurement process, ease of understanding and using the machine, the efficiency of the measurement process, and overall satisfaction with the experience. It aims to assess the user-friendliness and effectiveness of the machine from the subjects ' perspective.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The IP will be owned by the other company.